CLINICAL TRIAL: NCT06178081
Title: Effect of Non-Surgical Periodontal Treatment on Biomarker Levels in Smoker and Non-Smoker Periodontitis Patients
Brief Title: Effect of Non-Surgical Periodontal Treatment on Biomarker Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Burcu KARADUMAN, Proffesor, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2015-KAEK-79-23-08
Record Dates: First submitted 2023-12-04; First posted 2023-12-20 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2023-12

CONDITIONS: Healthy; Periodontitis
Keywords: periodontal therapy; biomarker; periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: Our study will include 50 people with periodontitis and 50 healthy periodontal patients (100 individuals in total), and these two groups will be divided into two as smokers and non-smokers. Clinical measurements (Plaque index, probing depth, gingival recession, clinical attachment level, bleeding on probing) salivary sample and gingival cerevicular fluid will be taken from all individuals at the beginning of the study. Non-surgical periodontal treatment will be applied to individuals with periodontitis, clinical measurements, saliva collection and gingival crevicular fluid will be repeated 12 weeks after the treatment. IL-39 analysis will be performed by ELISA in saliva and gingival crevicular fluid of individuals. IL-39 and cotinine levels will be examined to evaluate the effects of smoking before and after treatment in periodontal health and periodontitis.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clinical Healthy (Active Comparator): Clinical measurements (Plaque index, probing depth, gingival recession, clinical attachment level, bleeding on probing) salivary sample and gingival crevicular fluid will be taken from all individuals at the beginning of the study. IL-39 and cotinine levels will be examined to evaluate the effects of smoking before and after treatment in periodontal health and periodontitis. A pre-treatment saliva sample and gingival crevicular fluid will be collected from the clinically healthy group.
  Interventions: Other: Periodontal Healthy
- Periodontitis (Experimental): Non-surgical periodontal treatment will be applied to individuals with periodontitis, clinical measurements, saliva collection and gingival crevicular fluid will be repeated 12 weeks after the treatment. IL-39 analysis will be performed by ELISA in saliva and gingival crevicular fluid of individuals. IL-39 and cotinine levels will be examined to evaluate the effects of smoking before and after treatment in periodontal health and periodontitis. Clinical measurements (Plaque index, probing depth, gingival recession, clinical attachment level, bleeding on probing) and salivary sample will be taken from all individuals at the beginning of the study.
  Interventions: Other: Periodontal Healthy

INTERVENTIONS:
Other: Periodontal Healthy — Non surgical periodontal therapy
  Other Names: Periodontitis

SUMMARY:
Periodontitis is a destructive disease that follows untreated gingivitis and is characterized by gingival inflammation, clinical attachment loss, alveolar bone loss and periodontal pocket formation, increased tooth mobility and tooth loss. Although the primary etiological factor is microbial dental plaque, the host response plays an important role in the transition from periodontal health to disease. Smoking is a major risk factor for periodontitis and affects the formation and severity of the disease and healing after periodontal treatment by changing the host response to plaque. Proinflammatory and antiinflammatory cytokines have an important role in the pathogenesis of periodontal disease. Among these cytokines, interleukin (IL)-1β, IL-10 and currently IL-39 have been associated with periodontal disease. Further studies with post-treatment longitudinal evaluation are needed to elucidate the functions of IL-39 and its possible role in the pathogenesis of periodontal diseases. In this study, it was aimed to investigate the effects of non-surgical periodontal treatment on salivary and gingival crevicular fluid (GCF) IL-39, IL-1β and IL-10 levels in smokers and non-smokers with Stage 3 Grade B periodontitis and periodontally healthy individuals, both smokers and non-smokers. To the best of our knowledge, there is no study investigating the effects of non-surgical periodontal treatment and smoking on IL-39.

50 individuals with periodontitis and 50 periodontally healthy individuals (total 100 individuals) will be included in our study, and these two groups will be divided into two sub-groups as smokers and non-smokers. Clinical measurements (Plaque index, probing depth, gingival recession, clinical attachment level, bleeding on probing), saliva and GCF samples will be taken from all individuals at the beginning of the study. Non-surgical periodontal treatment will be performed in individuals with periodontitis. Saliva and GCF samples will be collected before treatment. The clinical measurements, saliva and GCF collection will be repeated 12 weeks after the treatment. The saliva and GCF levels of IL-39, IL-1β and IL-10 will be analyzed by ELISA. Cotinine levels will be examined to evaluate the effects of smoking before and after treatment in periodontal health and periodontitis.

With this study, we aimed to develop IL-39 diagnostic kits for the diagnosis of periodontal diseases, detection of disease activity, follow-up of response to treatment and healing.

ELIGIBILITY:
Inclusion Criteria:

* Periodontal healthy group
* Stage III Grade B and C Periodontitis Group
* To meet the above-mentioned periodontal health and disease criteria

Exclusion Criteria:

* Chronic alcohol use,
* Oral contraceptive use, pregnancy, pregnant,
* Last 6 months antibiotic or anti-inflammatory drug use,
* To have periodontal therapy in the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Examination of IL-39 levels of periodontal disease and clinically healthy | up to 1 year
  Examination of IL-39 levels, which are stated to be associated with periodontal disease, in gingival crevicular fluid and saliva samples obtained from individuals with periodontitis.

SECONDARY OUTCOMES:
Evaluation of the effect of non-surgical periodontal treatment on changes in IL-39 level. | up to 1 year
  Evaluation of the effect of non-surgical periodontal treatment on changes in IL-39 level.

OTHER OUTCOMES:
Comparison biomarkers of study groups. | up to 1 year
  Comparison of gingival crevicular fluid and saliva samples taken before treatment in individuals with periodontitis in terms of IL-39 levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided